CLINICAL TRIAL: NCT04090801
Title: Minoxidil in Treatment of Androgenetic Alopecia
Brief Title: Comparison of Topical Minoxidil 5% in Ethanol Plus Propylene Glycol Versus Minoxidil 5% in Ethanol Alone in Treatment of Women With Female Pattern Hair Loss
Acronym: FPHL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Abu El-Hamd, Assistant Professor of Dermatology, Venereology and Andrology Department, Faculty of Medicine, Sohag University, Egypt., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5/2015
Record Dates: First submitted 2019-08-30; First posted 2019-09-16 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Female Pattern Hair Loss
Keywords: Female pattern hair loss; Minoxidil.
MeSH Terms: interventions — Minoxidil; Ethanol; Propylene Glycol

STUDY DESIGN:
Intervention Model Description: This study will be to compare the efficacy of topical minoxidil 5% solution in ethanol plus 5% propylene glycol (PG), as a vehicle, versus 5% minoxidil in ethanol alone in treatment of women with FPHL.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The medications will be provided in bottles which will be identical in shape and color, and will be coded by a third party. Both patients and investigator will be blinded to the medication. Disclosure of the codes will be done, by a third party, at the end of the study.
Oversight: FDA-regulated Drug: No

ARMS (3):
- Topical minoxidil 5% in 90% ethanol and 5% propylene glycol (Active Comparator): Group A applied topical minoxidil 5% in 90% ethanol and 5% propylene glycol
  Interventions: Drug: Topical minoxidil 5% in 90% ethanol and 5% propylene glycol
- Topical minoxidil 5% in pure ethanol alone (Active Comparator): Group B applied topical minoxidil 5% in pure ethanol alone
  Interventions: Drug: Topical minoxidil 5% in pure ethanol alone
- Placebo (Placebo Comparator): Group C applied pure ethanol (placebo)
  Interventions: Other: Placebo (Ethanol)

INTERVENTIONS:
Drug: Topical minoxidil 5% in 90% ethanol and 5% propylene glycol
  Other Names: Topical minoxidil 5% with 90% ethanol and 5% propylene glycol
  Arms: Topical minoxidil 5% in 90% ethanol and 5% propylene glycol
Drug: Topical minoxidil 5% in pure ethanol alone — The treatment will be continued twice daily.for six months with regular visits at 3 months intervals.
  Other Names: Topical minoxidil 5%
  Arms: Topical minoxidil 5% in pure ethanol alone
Other: Placebo (Ethanol) — The treatment will be continued twice daily.for six months with regular visits at 3 months intervals.
  Arms: Placebo

SUMMARY:
The study will be included 60 women with FPHL. The diagnosis of FPHL will be established by clinical (Ludwig classification) and trichoscopic evaluation of frontal and occipital regions of the scalp.

DETAILED DESCRIPTION:
Enrolled women will be randomly assigned into 3 treatment groups: group A will apply topical minoxidil 5% in 90% ethanol and 5% propylene glycol, group B will apply topical minoxidil 5% in pure ethanol alone and group C will apply pure ethanol (placebo) twice daily.

The treatment will be continued for six months with regular visits at 3 months intervals.

The medications will be provided in bottles which were identical in shape and color, and were coded by a third party.

Both patients and investigator will be blinded to the medication. Disclosure of the codes will be done, by a third party, at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* FPHL

Exclusion Criteria:

* No

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05-30 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Ludwig scale grading system | 0-6 months
  The 3 grades will be defined. Grade 1, (Thinning of hair is seen mainly over the anterior part of the crown with minimal widening of the parting width). Grade 2, (Thinning of the crown becomes more evident because of an increase in the number of thin and short hairs). Grade 3, (The crown becomes almost total bald, but the frontal hair line is still maintained).
Trichoscopic examination of the hairs at frontal and occipital regions of the scalp. | 0-6 months
  It will be evaluated signs of hair changes such as hair diameter diversity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abu El-Hamd, MD, Principal Investigator — Faculty of Medicine, Sohag University, Egypt.

IPD SHARING:
Plan to Share IPD: No